CLINICAL TRIAL: NCT00078208
Title: Exhaled Breath Condensate as a Measurement of Airway Inflammation in Children With Asthma
Brief Title: Exhaled Breath Condensate as a Measure of Airway Inflammation in Children With Asthma
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040126; 04-I-0126
Record Dates: First submitted 2004-02-19; First posted 2004-02-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-08-19

CONDITIONS: Asthma
Keywords: Pediatric; Non-Invasive; Anti-Inflammatory; pH; Mediators; Asthma; Childhood Asthma; Healthy Volunteer; HV
MeSH Terms: conditions — Asthma

SUMMARY:
This study will evaluate the usefulness of a new procedure for evaluating asthma in children. The method measures the pH (a measure of acidity and alkalinity) of exhaled breath condensate (water vapor created by the lungs). The condensate contains products of the lungs that may be associated with lung inflammation. Investigators will determine if the pH of the exhaled breath condensate correlates well with known asthma indicators, such as number of hospitalizations, school absenteeism, use of rescue medication, and others. Test results will be compared with findings from healthy normal volunteers. No experimental treatments or medicines are used in this study. Patients who require treatment for their asthma will receive standard care with medicines approved by the Food and Drug Administration and used widely in the United States.

Children with asthma and healthy normal volunteers between 6 and 17 years of age may be eligible for this study. You must complete the study before your 18th birthday. Candidates are screened with a medical history and physical examination.

Children with asthma undergo the following tests and procedures over six clinic visits, including an initial visit and follow-up visits at 4-8 weeks, 3, 6, 9, and 12 months:

* Blood draw in children over 6 years of age. Medications are available to decrease the pain associated with blood drawing.(initial visit)
* Allergen skin testing: Drops of up to 16 allergens are placed on the arm. The skin under each drop is scratched and the area is observed for an allergic reaction. (4- 8-week follow-up visit)
* Expired nitric oxide testing: The child breathes into a balloon to collect a portion of the gases exhaled form the lungs. This test measures the amount of nitric oxide, which correlates with bronchial inflammation. (all visits)
* Exhaled breath condensate: The child breathes into a plastic tube surrounded by a cold metal sleeve for 10 to 15 minutes. The water vapor created by the lungs (the same vapor that forms when breathing outside on a cold day) is collected and the pH measured. (all visits)
* Pulmonary (lung) function test: The child blows very hard into a tube attached to a machine to measure the airflow from the child's lungs. This test measures airflow from the lungs. (all visits) The children are given small plastic device called a peak flow meter - a device used to measure lung function - to use at home. Children whose lung function is less than 80% of the predicted value for their age may be given medicine to see if their lung function improves.
* Review of the patient's symptoms, sick days, medicines or actions taken to get over the illness; review of peak flow reports; and review of action plan. (3-, 6-, 9-, and 12-month visits)

Healthy controls will have the expired nitric oxide test, exhaled breath condensate test, and pulmonary function test at each visit at the initial and over two additional visits scheduled 6 months apart.

DETAILED DESCRIPTION:
The onset of asthma is often during childhood, and when the child is atopic, it is more likely to persist into adulthood. Diseases such as asthma have a higher prevalence in childhood; and management that alters the morbidity of allergic disease in children may impact disease outcomes in future years.

Asthma is the most prevalent chronic disease in childhood and accounts for the highest rate of hospitalizations in the ages between 0-4 years. Unfortunately, there are few noninvasive objective measurements of pulmonary health in children. Current techniques include determination of peak flow, spirometry, and measurement of nitric oxide (NO). Bronchial inflammation is a central feature of asthma and anti-inflammatory therapy is the mainstay of treatment. Expired NO (eNO) has been shown to correlate with bronchial inflammation. However, the collection of NO has only been available in research settings due to the limitations of collection and analysis. In contrast, exhaled breath condensate (EBC) is easily obtained and pH analysis technically simple.

Determination of pH in EBC is a novel, non-invasive technique in clinical study as a means to evaluate the severity of pulmonary inflammation. In the protocol described, we will evaluate the utility of EBC in the measurement of airway disease in 60 children with asthma and compare them to 30 healthy cohorts in the same age range. We will determine if EBC pH is reflective of the degree of morbidity in children by correlating measurements with known parameters of disease including: 1) number of hospitalizations, 2) absenteeism from school, 3) number of asthma exacerbations, 4) loss of work days (if applicable), 5) extent of rescue medication usage, 6) spirometry to evaluate obstruction, and 7) NO as a measurement of inflammation.

Subjects will be evaluated and then categorized based on the National Asthma Education and Prevention Program (NAEPP) guidelines. We will measure the pH from EBC in children age 6 to less than 18 years of age and compare findings to clinical data, spirometry, and expired NO. In this way, we will determine if EBC is a potentially useful non-invasive measurement of airway disease. It is hoped that measurements of EBC will be helpful in identifying those children in which the addition of an anti-inflammatory medication is appropriate. We will also attempt to measure inflammatory mediators to determine if they can be used to assess inflammation.

This method may also be useful in detecting airway inflammation due to an infectious agent before a systemic reaction (fever, respiratory distress, or cough) is apparent in children with various immunodeficiency diseases such as chronic granulomatous disease (CGD), recurrent respiratory infections without a defined host defect (RIND), or Job's syndrome.

We will recruit 30 healthy control children in the same age range to compare the EBC pH values in children without allergic or other chronic pulmonary diseases. In addition, we will recruit 30 children (10 in each group) with CGD, RIND, and Job's to compare exhaled breath condensate pH and exhaled nitric oxide values to those from children with allergic airway inflammation to determine if these methods are useful for early diagnosis of infectious airway inflammation.

ELIGIBILITY:
* INCLUSION CRITERIA:

ASTHMA:

Children ages 5 to less than 18 years at the time he or she is expected to complete the protocol with asthma. One or more of the following criteria will qualify for inclusion:

Doctor diagnosed asthma.

Chronic cough, worse particularly at night for greater than one month.

Recurrent wheezing during the past 6 months.

Symptoms of difficulty breathing occurring concurrently or worsened by, exercise, infection, animals, smoke, pollen or strong emotional expression.

Medical care for treatment of respiratory symptoms consistent with asthma.

Reversible (greater than or equal to 12%) airflow obstruction after an inhaled short-acting beta2-agonist.

HEALTHY CONTROL:

Children between the ages of 5 and less than 18 years at the time he or she is expected to complete the protocol.

Subject (asthma or healthy control) has a non-NIH physician who provides routine and emergency care. When available, permission for access of medical records and pharmacy records will be obtained for subjects with asthma.

SUBJECT WITH IMMUNODEFICIENCY:

Children between the ages of 5 and less than 18 at the time he or she is expected to complete the protocol.

Doctor diagnosed immunodeficiency (CGD, Job's, RIND).

EXCLUSION CRITERIA:

Unacceptably poor compliance, which in the opinion of the investigator, would interfere with one's ability to study or provide medical care for the subject.

Any major illness or condition that, in the opinion of the principal investigator, may interfere with the subject's ability to comply with the conditions of participation in the study:

Latex allergy

Current tobacco use.

URI symptoms in the 4 weeks prior to EBC collection.

Any condition that, in the opinion of their primary physician, would affect your child's participation in the study.

HIV negative by history.

HEALTHY CONTROL:

Asthma or allergic rhinitis.

Chronic pulmonary disease.

URI symptoms in the 4 weeks prior to EBC collection.

Chronic corticosteroid therapy (daily or every other day dosing for greater than 14 days).

Current tobacco use.

HIV negative by history.

History of latex allergy.

PATIENTS WITH IMMUNODEFICIENCY:

Chronic or prophylactic antibiotics.

Diagnosis of asthma.

Must be off antibiotics for 2 days.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2004-02-18; Study Completion 2010-08-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Smith DH, Malone DC, Lawson KA, Okamoto LJ, Battista C, Saunders WB. A national estimate of the economic costs of asthma. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):787-93. doi: 10.1164/ajrccm.156.3.9611072. PMID 9309994
- [Background] Newacheck PW, Taylor WR. Childhood chronic illness: prevalence, severity, and impact. Am J Public Health. 1992 Mar;82(3):364-71. doi: 10.2105/ajph.82.3.364. PMID 1536351
- [Background] Halfon N, Newacheck PW. Childhood asthma and poverty: differential impacts and utilization of health services. Pediatrics. 1993 Jan;91(1):56-61. PMID 8416505